CLINICAL TRIAL: NCT04604639
Title: Do Patients Suffering an Out-of-hospital Cardiac Arrest Present to the Ambulance Service With Symptoms in the Preceeding 48hrs?
Brief Title: Do Patients Suffering a Cardiac Arrest Present to the Ambulance Service With Symptoms in the Preceeding 48hrs?
Status: Completed | Type: Observational
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: South Central Ambulance Service NHS Foundation Trust (Unknown)
Responsible Party: Sponsor
Other Study IDs: 3724/18
Record Dates: First submitted 2020-10-21; First posted 2020-10-27 (Actual); Last update posted 2022-04-13 (Actual); Status verified 2020-02

CONDITIONS: Cardiac Arrest
Keywords: Cardiac arrest; Ambulance; Triage; Deterioration
MeSH Terms: conditions — Heart Arrest

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Out-of-hospital cardiac arrest: Patients suffering an out-of-hospital cardiac arrest to who the ambulance service was requested to attend.
  Interventions: Diagnostic Test: NEWS2 score

INTERVENTIONS:
Diagnostic Test: NEWS2 score — Patients seen by ambulance crews within the preceeding 48 hrs of their cardiac arrest will have a NEWS2 score performed to assess the level of physiological deterioration at the time of thei intial assessment.

SUMMARY:
A cardiac arrest is often preceeded by a varying period of physiological deterioration which if acted upon may prevent the cardiac arrest. We aim to review patients presenting to the ambulance service with cardiac arrest so see if they had contacted the ambulance service in the preceeding 48 hrs to understand if warning symptoms were missed or not acted upon appropriately.

DETAILED DESCRIPTION:
The UK ambulance services are called to attend 60,000 out-of-hospital cardiac arrests (OHCA) each year. Hospital studies have shown that many patients who suffer an in-hospital cardiac arrest (IHCA) have been deteriorating for the preceeding 48 hrs and suggest that many IHCA are potentially avoidable if this deterioration is identified and actued on promptly. No similar study has been performed to see if patients suffering OHCA have also presented with warning signs in the preceeding 48 hrs that were overlooked.

ELIGIBILITY:
Inclusion Criteria:

• All patients seen by SCAS ambulance crews and suffering a cardiac arrest within the following 48 hrs

Exclusion Criteria:

• None

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Study Population: All patients calling for an emergency ambulance in the South Central Ambulance Service region, where an emergency ambulnace was dispatched and a patient intervention occurred.
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-02-01 (Actual); Primary Completion 2020-02-19 (Actual); Study Completion 2020-02-20 (Actual)

PRIMARY OUTCOMES:
Out-of-hospital cardiac arrest | 48 hours
  Cardiac arrest following ambulance assessment

CONTACTS AND LOCATIONS:
Overall Officials: Charles D Deakin, MD, Principal Investigator — Divisional Medical Director
Locations (1):
- South Central Ambulance Service, Otterbourne, Hampshire, United Kingdom